CLINICAL TRIAL: NCT02467959
Title: Diagnostic Accuracy and Clinic Utility of Bedside Ultrasonography Performed by Emergency Physicians in Suspected Acute Appendicitis
Brief Title: Diagnostic Accuracy of Emergency Physician Performed Bedside Ultrasound in Suspected Acute Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, faruk güngör, MD, Antalya Training and Research Hospital
Other Study IDs: AntalyaTRH04
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Acute Abdomen; Acute Appendicitis
Keywords: emergency ultrasound; acute appendicitis; bedside ultrasound
MeSH Terms: conditions — Abdomen, Acute; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound: Ultrasound evaluation

SUMMARY:
The aim of the study is to evaluate the diagnostic yield and accuracy of bedside emergency physician performed ultrasound in the diagnosis of acute appendicitis.

DETAILED DESCRIPTION:
Emergency physician (EP) performed bedside ultrasound is cost effective, repeatable and especially useful in the diagnosis of life treating conditions such as aortic dissection, traumatic bleedings. While abdominal pain is a common complaint in the emergency department and accurate diagnosis of its etiology may affect the patient's outcome, the accuracy and the diagnostic yield of bedside EP performed ultrasound is not well established. The diagnosis of a patient presented to emergency department with right lower abdominal pain is generally problematic and physician has to exclude acute surgical reasons such as acute appendicitis.

In this study, patients who are suspicious to have acute appendicitis base on their clinical findings will be included. EP will record his diagnosis and then patient will undergo emergency physician performed ultrasound. After ultrasound EP will fill the study form according to US findings and record his diagnosis once again.

At the end of the study the investigators evaluate and compare the radiology performed US reports and if there is operational biopsy results with the EP's pre- and post ultrasound diagnosis to estimate the diagnostic yield and accuracy of bedside emergency physician performed ultrasound in the diagnosis of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with the complaint of right lower abdominal pain
* Suspected acute appendicitis

Exclusion Criteria:

* Flank pain
* Previous appendectomy
* Pregnancy
* Unstable vital signs
* Frank peritonitis
* US performed before EP's examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age presented to emergency department with the complaint of right lower abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of emergency physician performed bedside ultrasound in diagnosing of acute appendicitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: faruk güngör, md, Study Chair — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Emergency, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Hussain S, Rahman A, Abbasi T, Aziz T. Diagnostic accuracy of ultrasonography in acute appendicitis. J Ayub Med Coll Abbottabad. 2014 Jan-Mar;26(1):12-7. PMID 25358207
- [Result] Lam SH, Grippo A, Kerwin C, Konicki PJ, Goodwine D, Lambert MJ. Bedside ultrasonography as an adjunct to routine evaluation of acute appendicitis in the emergency department. West J Emerg Med. 2014 Nov;15(7):808-15. doi: 10.5811/westjem.2014.9.21491. Epub 2014 Sep 18. PMID 25493122